CLINICAL TRIAL: NCT02863510
Title: Renal Sympathetic Denervation in Moderate to Severe Chronic Kidney Disease Using a Novel Non-iodinated Contrast Free Protocol
Brief Title: Renal Sympathetic Denervation in Moderate to Severe Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart of England NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012138RN
Record Dates: First submitted 2016-02-12; First posted 2016-08-11 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Carbon dioxide angiography; Renal sympathetic denervation; Uncontrolled hypertension; Chronic kidney disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation (Experimental): Participation receiving renal sympathetic denervation
  Interventions: Device: Renal Sympathetic Denervation

INTERVENTIONS:
Device: Renal Sympathetic Denervation — Renal sympathetic denervation is a minimally invasive, endovascular catheter-based procedure using radiofrequency ablation of sympathetic nerves located in the walls of renal arteries, aimed at treating treatment-resistant hypertension.

SUMMARY:
A pilot, single-center, prospective, interventional study. The objective is to demonstrate that catheter-based renal denervation using carbon dioxide renal angiography in patients with moderate to severe chronic kidney disease can be performed for treatment of uncontrolled hypertension.

DETAILED DESCRIPTION:
Renal sympathetic denervation has been shown to be safe and effective in patients with uncontrolled hypertension and estimated Glomerular Filtration Rate (eGFR)>45 mL/min per 1•73 m². However, the safety and efficacy of this has not been studied in patients with more severe renal impairment. The investigators aim to examine safety and efficacy of renal denervation (RDN) in patients with eGFR between 44 and 15 ml/min/1.73 m2 (CKD 3b & 4) in a pilot study which may be a precursor of a large observational study in the future. Moreover, the current imaging protocol and procedure protocol for renal sympathetic denervation requires the use of iodinated contrast, which can have deleterious effects on renal function. The investigators have a proven track record for the use of carbon dioxide angiography in renal artery intervention. The investigators would like to use carbon dioxide angiography in this study to minimize contrast induced deterioration in renal function in this cohort which may again be a precursor of a farther larger study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years with a clinic systolic blood pressure of 140 mm Hg or more despite compliance with three or more antihypertensive drugs,
* eGFR<45 and >15 mL/min per 1.73 m².

Exclusion Criteria:

* eGFR <15 mL/min per 1.73 m²,
* Type 1 diabetes,
* Substantial stenotic valvular heart disease,
* Pregnancy or planned pregnancy during the study,
* A history of myocardial infarction, unstable angina, or cerebrovascular accident in the previous 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Estimated glomerular filtration rate from baseline to 7 days and 30 days | at baseline, 7days and 30 days
  Change in eGFR from baseline to 7 days and 1 month as measure of safety in terms of kidney function

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate from baseline to 7 days, 1, 3, and 6 months | at baseline, 7 days, 1, 3, and 6 months
  Change in kidney function from baseline to 7 days, 1, 3, and 6 months
Change in proteinuria (albumin:creatinine ratio) from baseline to at 1, 3, and 6 months. | at baseline, 1, 3, and 6 months
  Change in proteinuria (albumin:creatinine ratio) from baseline to at 1, 3, and 6 months.
Change in mean daytime ambulatory blood pressure on 24 hour monitoring from baseline to 6 months | at baseline and 6 months
  Change in mean daytime ambulatory blood pressure on 24 hour monitoring from baseline to 6 months
Change in office blood pressure from baseline to 1,3, and 6 months | at baseline, 1, 3, and 6 months
  Change in office BP from baseline to 1,3, and 6 months for efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Indranil Dasgupta, DM, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Heart of England NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No